CLINICAL TRIAL: NCT00092950
Title: A Pilot Study of a Three Month Intervention for Increasing Physical Activity in Sedentary Women at Risk for Breast Cancer
Brief Title: Exercise in Women at Risk for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Giuseppe Giaccone, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040276; 04-C-0276; NCT00095849 (obsolete NCT alias)
Record Dates: First submitted 2004-09-24; First posted 2004-09-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-28

CONDITIONS: Breast Neoplasms
Keywords: Exercise; Pedometer; Physician Prescription; Biomarkers; Compliance; Breast Cancer Survivor; Breast Cancer Risk
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Patient Compliance | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical activity

SUMMARY:
This 2-part study will examine how much exercise people usually do in the course of their daily lives and how two different types of exercise-stretching and walking-affect the amount of fat in the body and certain hormones in the blood. It will also examine whether exercise can be increased by physician counseling with and without the use of a pedometer, and if exercising changes levels of stress, anxiety, and depression.

Breast cancer survivors and women at high risk for breast cancer who are between 18 and 75 years of age and who exercise less than 3 times per week may be eligible for this study. Candidates are screened with a medical history and physical examination, and their endurance and flexibility are tested by stretching exercises and by a 6-minute walk or run.

All participants complete study Part 1. Those who are eligible may also participate in Part 2.

* Part 1: Subjects wear a pedometer (a small device that measures the number of steps taken) on their waistband during all waking hours for 1 week without changing their usual level of activity. Depending on their level of activity, subjects may be invited to participate in Part 2 of the study.
* Part 2: Subjects are placed in either a walking group or a stretching group for 12 weeks. At the end of the 12-week period, those in the walking group are offered participation in the stretching group, and those in the stretching group are offered participation in the walking group.

Walking group participants wear a pedometer every day for 12 weeks. They are asked to gradually increase the number of steps they take each day, to keep a record of their daily step count, and to report periodically to the study staff on their progress. For 1 week during the study, participants also wear a device called an accelerometer that is used to verify the accuracy of the pedometer step counts.

Stretching group participants follow a program of stretching exercises for 12 weeks, with their progress monitored periodically by staff. During week 12, participants wear a pedometer and accelerometer.

All Part 2 participants also have the following tests and procedures:

* Blood draw: collected at the beginning and end of the study to test for certain hormones and HDL cholesterol levels.
* Questionnaires: about stress, anxiety, and depression levels; these are completed at the beginning and end of the study, and a detailed questionnaire about diet is completed at home or during a clinic visit.
* Body composition measurement: A "bioelectrical impedance" test, which measures body fat, is done at the beginning and end of the study. For this test, the subject lies on an examining table and a small electrical current is passed through electrodes placed on one hand and one foot. Although a small electrical current is used, this test is not painful.
* Endurance and flexibility testing: At the end of the study, participants repeat the 6-minute walk or run endurance test and the stretching flexibility test performed at screening.

DETAILED DESCRIPTION:
Background:

Evidence suggests that high levels of physical activity can decrease breast cancer risk.

Physical activity could therefore represent a viable breast cancer prevention strategy.

In order to study the effect of physical activity on breast cancer risk, we must first develop feasible and efficacious physical activity interventions.

Objectives:

Primary:

To determine the rate of compliance with a physical activity intervention using a pedometer, a physician prescription, and a motivational booklet.

To determine whether this intervention is more effective than a control of stretching exercises at increasing physical activity.

Secondary:

To determine whether physical activity as measured by a pedometer correlates with other measures of physical activity.

To assess the effect of the physical activity intervention on serum biomarkers, quality of life, functional capacity and body composition.

To examine long-term compliance with a program of increased physical activity and assess post program exercise motivation and adherence.

Eligibility:

Eligible patients are women age 18-75 who meet one of the following criteria:

History of breast cancer without evidence of recurrent disease.

Gail model 5 year risk greater than 1.7%.

Claus model lifetime risk greater than 20%.

History of appropriately treated DCIS.

History of high risk lesion on breast biopsy (ADH, ALH, LCIS).

Known or suspected BRCA1 or BRCA2 mutation.

Patients must be sedentary at baseline and must be medically fit to exercise.

Design:

This is a randomized pilot study designed to assess the feasibility of a physical activity intervention in breast cancer survivors and women at high risk for breast cancer.

Stage I: Patients undergo a baseline activity evaluation for one week which involves wearing a sealed pedometer - those that have an average daily step count of less than 5,000 steps are eligible for randomization.

Stage II: Patients are assigned to either a walking intervention, (including a pedometer, a physician exercise prescription with a final goal of walking 10,000 steps per day, and a motivational booklet) or a control of stretching exercise for a period of 12 weeks.

Biomarkers, functional capacity, body composition and diet are assessed at the beginning and end of study.

This study plans to randomize 80 subjects, and has a greater than 90% power to detect a mean increase of 3,000 steps per day in intervention subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will enroll 40 breast cancer survivors and 40 women at high risk for breast cancer. All participants must fulfill the following criteria:

Age 18 to 75.

Sedentary at baseline, as defined by a weekly leisure-time activity score of 15 or less on the Godin Leisure-Time Exercise Questionnaire. This cutoff is equivalent to engaging in moderate activity less than 3 times a week.

Ability to complete all study questionnaires, or a willing friend or family member who will assist in questionnaire completion.

ECOG performance status 0-1.

Ability to successfully perform the level of physical activity prescribed by the protocol, as assessed by the Physical Activity Readiness Questionnaire (PAR-Q).

Any participant who answers yes to any of the questions in this screening tool will undergo medical evaluation at the Clinical Center, as appropriate, prior to enrolling on the study.

Cardiac risk will be assessed after a complete history and physical exam, and will be determined by the examining physician. Only patients who are felt to be increased cardiac risk will have an EKG performed. This will include patients who answer yes to any of the questions on the PAR-Q that assess cardiac risk (#1,2,3,4,6). Patients with worrisome EKG findings or findings in the history or physical exam that warrant further work-up in the opinion of the health care provider will be referred to the cardiology consult service, or if non-urgent, will be referred back to their source of regular medical care for clearance prior to enrolling on the study.

If history of cancer (other than invasive breast cancer, squamous or basal cell skin cancers), subject must have no evidence of disease at time of enrollment AND no history of cancer directed treatment in the 2 years preceding enrollment.

Breast cancer survivors:

Eligible breast cancer survivors will be women with a documented history of Stage I, II or III invasive breast cancer who are at least two months from the completion of their primary therapy, including surgery, radiation and chemotherapy. Current use of hormonal therapy such as tamoxifen or aromatase inhibitors, will be permitted, however subjects must have completed 2 months of hormonal therapy prior to beginning the study in order to achieve steady state.

Women at high risk for breast cancer:

Women will be considered at high risk for developing breast cancer if they fulfill one of the following criteria:

A Gail model risk of greater than or equal to1.7 percent over 5 years from study entry or a Claus model lifetime risk of greater than 20 percent.

Lobular neoplasia.

Atypical ductal hyperplasia.

Ductal carcinoma in situ (DCIS) that has been previously treated. Patients must be at least 2 months from completion of primary therapy, and if treated with hormonal therapy, they must have completed at least two months of hormonal therapy.

Deleterious mutations in BRCA-1 or 2 OR A priori risk assessment of 20 percent chance or greater of carrying a BRCA1/2 gene mutation. The BRCAPRO model (109) will be used to assess this risk.

EXCLUSION CRITERIA:

Currently pregnant or planning to become pregnant during the study period. Pregnancy will be assessed in women of childbearing potential prior to enrolling in stage II of the study. Postmenopausal women and women who have had a previous hysterectomy, oophorectomy or tubal ligation will not be required to undergo a pregnancy test.

Uncontrolled intercurrent illness, including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recent myocardial infarction or stroke, or psychiatric illness/social situations that would limit compliance with study requirements.

Physical conditions that preclude the amount of daily walking prescribed by the protocol (e.g., severe arthritis, use of a walker or cane, wheelchair-bound, etc.).

Medical or psychiatric disorder which would, in the opinion of the Principal Investigator, render the subject unable to provide informed consent.

Patients with metastatic or recurrent disease will be excluded because of difficulty interpreting results in the context of women with a disease burden and/or on chemotherapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-09-23; Primary Completion 2009-12-07 (Actual); Study Completion 2009-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Freedman AN, Graubard BI, Rao SR, McCaskill-Stevens W, Ballard-Barbash R, Gail MH. Estimates of the number of US women who could benefit from tamoxifen for breast cancer chemoprevention. J Natl Cancer Inst. 2003 Apr 2;95(7):526-32. doi: 10.1093/jnci/95.7.526. PMID 12671020
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446